CLINICAL TRIAL: NCT07141316
Title: Effects of Blood Flow Restriction Combined With Electrostimulation After Knee Arthroplasty: Randomized Controlled Trial
Brief Title: Effects of Blood Flow Restriction Combined With Electrostimulation After Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFR01
Record Dates: First submitted 2025-08-04; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Osteo Arthritis Knee
Keywords: Blood Flow Restriction, Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction and Electrostimulation (GEL) (Experimental): For six working days, starting from the third day after surgery, he will perform 30 minutes of blood flow restriction once a day during electrostimulation of the quadriceps of the operated limb.
  Interventions: Device: Blood flow restriction combined with electrostimulation.
- Electrostimulation alone (GST) (No Intervention): For six working days, starting from the third day after surgery, he will perform 30 minutes of electrostimulation of the quadriceps of the operated limb once a day

INTERVENTIONS:
Device: Blood flow restriction combined with electrostimulation. — Participants will perform 30 minutes of blood flow restriction once a day during electrostimulation of the quadriceps of the operated limb.
  Arms: Blood flow restriction and Electrostimulation (GEL)

SUMMARY:
The goal of this clinical trial is to learn whether blood flow restriction (BFR) combined with electrostimulation (ES) can improve the postoperative course of patients undergoing total knee arthroplasty. The main questions it aims to answer are:

Immediately after surgery, do BFR combined with ES increase quadriceps strength? Do they also improve the functional abilities of patients? Researchers will compare BFR combined with ES to ES alone, to see if there are differences.

Participants will carry out a daily session of BFR+ ES or ES alone for six working days after surgery

DETAILED DESCRIPTION:
Blood flow restriction (BFR) is an innovative treatment technique that involves the application of controlled pressure, through a special sleeve, to partially limit arterial flow and completely prevent venous outflow in the active muscles during exercise.

This approach is based on a hemodynamic modulation that induces a hypoxic environment at the muscle level, favoring the activation of metabolic processes and cellular mechanisms responsible for positive adaptations, such as the increase in protein synthesis, the promotion of muscle hypertrophy, aerobic capacity and the management of pain perception.

In rehabilitation, blood flow restriction treatment has been recognized as an effective strategy to promote functional recovery, offering benefits comparable to those of traditional treatment with high loads. This methodology is particularly useful in contexts where the use of high loads is contraindicated, such as in patients with orthopaedic limitations, with muscle weakness or undergoing surgery because it induces significant muscle adaptation even with low loads. The latest evidence indicates that reduced Limb occlusion pressures (LOP) (40% of blood pressure) achieve similar benefits to high pressures (80%) and are appreciated by patients. In the middle-aged and elderly population, the efficacy of BFR has been widely demonstrated but the studies that have investigated its effects on patients undergoing Knee Arthroplasty (KA) are few, of poor quality and carried out in the advanced rehabilitation phase. Patients undergoing KA at the "Città di Pavia" University Hospital, from the first post-operative day, perform a standard rehabilitation program including: passive mobilization, assisted active exercises, indirect electrostimulation and gait re-education. Although the results are positive, in the first few days, there are cases in which problems such as loss of muscle strength and functionality and persistence of pain occur; these sequelae are in agreement with the most recent literature.

Based on the rationale, the study aims to evaluate, in a group of patients undergoing KA, the short-term effects of electrostimulation combined with BFR and compare them with those of a group that will carry out the standard treatment. The treatment steps will be as follows:

I. positioning of electrodes for electrostimulation on the quadriceps of the operated limb; II. application of the pneumatic band to the root of the thigh and LOP setting; III. programmazione dei parametri della BFR (LOP, 50%) (Occlusion time, 6 periods of 4 minutes of occlusion and 1 minutes of rest); IV. simultaneous start-up of the two devices.

ELIGIBILITY:
Inclusion Criteria:

* Elective knee arthroplasty surgery

Exclusion Criteria:

* obesity (body mass index equal to or greater than 30 Kg/m2);
* concomitant orthopaedic or neurological pathologies (other than the pathology for which arthroprosthesis has been indicated) that modify walking capacity;
* pathologies that modify the balance (neurological and/or vestibular);
* contraindications to the use of medical equipment used in the practice;
* inability to understand and sign informed consent.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Maximum quadriceps strength of the operated limb | From the second to the tenth day post surgery.
  Maximum quadriceps strength, measured with a dynamometer and expressed in kilograms

SECONDARY OUTCOMES:
Functional Capacities | From the second to the tenth day post surgery.
  Timed Up and Go test ( seconds) and the 30 Seconds Chair Stand test (number of repetitions) will performed.
Functional Strength | From the second to the tenth day post surgery.
  30 Seconds Chair Stand test (number of repetitions)
Walking autonomy | From the second to the tenth day post surgery.
  20 meters walking test (seconds)

CONTACTS AND LOCATIONS:
Overall Officials: luca Marin, PhD, Principal Investigator — University of Pavia
Locations (1):
- Istituto di Cura "Città di Pavia", Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
On justified request and in anonymised form.
Supporting Information: Analytic Code
Time Frame: From the publication of the study (start date) for five years (end date).
Access Criteria: Only researchers who request it for a justified reason will be able to access the data in anonymized form

REFERENCES:
- [Result] Praetorius A. [Blood flow restriction training (BFRT) in patients before and after total knee arthroplasty]. Orthopadie (Heidelb). 2024 Nov;53(11):853-857. doi: 10.1007/s00132-024-04543-1. Epub 2024 Aug 9. German. PMID 39120683
- [Result] Conference Proceedings for the 10th Annual Meeting of Arthroplasty Society in Asia (ASIA), 26th Annual Meeting of the Thai Hip and Knee Society (THKS), and the 16th Annual Meeting of the ASEAN Arthroplasty Association (AAA). Arthroplasty. 2024 Dec 20;6(Suppl 1):62. doi: 10.1186/s42836-024-00286-8. No abstract available. PMID 39702276
- [Result] Wengle L, Migliorini F, Leroux T, Chahal J, Theodoropoulos J, Betsch M. The Effects of Blood Flow Restriction in Patients Undergoing Knee Surgery: A Systematic Review and Meta-analysis. Am J Sports Med. 2022 Aug;50(10):2824-2833. doi: 10.1177/03635465211027296. Epub 2021 Aug 18. PMID 34406084
- [Result] De Renty C, Forelli F, Mazeas J, Kakavas G, Hewett TE, Korakakis V. Knee Loading With Blood Flow Restriction Can Enhance Recovery After Total Knee Arthroplasty. Cureus. 2023 Apr 20;15(4):e37895. doi: 10.7759/cureus.37895. eCollection 2023 Apr. PMID 37214015
- [Result] Zhang T, Wang X, Wang J. Effect of blood flow restriction combined with low-intensity training on the lower limbs muscle strength and function in older adults: A meta-analysis. Exp Gerontol. 2022 Jul;164:111827. doi: 10.1016/j.exger.2022.111827. Epub 2022 May 1. PMID 35508279
- [Result] Chang H, Yao M, Chen B, Qi Y, Zhang J. Effects of Blood Flow Restriction Combined with Low-Intensity Resistance Training on Lower-Limb Muscle Strength and Mass in Post-Middle-Aged Adults: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2022 Nov 25;19(23):15691. doi: 10.3390/ijerph192315691. PMID 36497769
- [Result] Das A, Paton B. Is There a Minimum Effective Dose for Vascular Occlusion During Blood Flow Restriction Training? Front Physiol. 2022 Apr 8;13:838115. doi: 10.3389/fphys.2022.838115. eCollection 2022. PMID 35464074
- [Result] Freitas EDS, Miller RM, Heishman AD, Ferreira-Junior JB, Araujo JP, Bemben MG. Acute Physiological Responses to Resistance Exercise With Continuous Versus Intermittent Blood Flow Restriction: A Randomized Controlled Trial. Front Physiol. 2020 Mar 17;11:132. doi: 10.3389/fphys.2020.00132. eCollection 2020. PMID 32256374
- [Result] Barber-Westin S, Noyes FR. Blood Flow-Restricted Training for Lower Extremity Muscle Weakness due to Knee Pathology: A Systematic Review. Sports Health. 2019 Jan/Feb;11(1):69-83. doi: 10.1177/1941738118811337. Epub 2018 Nov 26. PMID 30475660
- [Result] Loenneke JP, Abe T, Wilson JM, Thiebaud RS, Fahs CA, Rossow LM, Bemben MG. Blood flow restriction: an evidence based progressive model (Review). Acta Physiol Hung. 2012 Sep;99(3):235-50. doi: 10.1556/APhysiol.99.2012.3.1. PMID 22982712
- [Result] Bielitzki R, Behrendt T, Behrens M, Schega L. Time to Save Time: Beneficial Effects of Blood Flow Restriction Training and the Need to Quantify the Time Potentially Saved by Its Application During Musculoskeletal Rehabilitation. Phys Ther. 2021 Oct 1;101(10):pzab172. doi: 10.1093/ptj/pzab172. PMID 34228788
- [Result] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Result] A. K. Sandilya, D. Kashyap, A. Arunmozhi, M. Wadhwa, e V. Verma, "The importance of Blood Flow Restriction Training (BFRT) in Physiotherapy: A Review of Literature", J. Reatt. Ther. Dev. Divers., ago. 2023, doi: 10.53555/jrtdd.v6i8s.2643.
- [Result] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Result] Xia B, Di Chen, Zhang J, Hu S, Jin H, Tong P. Osteoarthritis pathogenesis: a review of molecular mechanisms. Calcif Tissue Int. 2014 Dec;95(6):495-505. doi: 10.1007/s00223-014-9917-9. Epub 2014 Oct 14. PMID 25311420
- [Result] Litwic A, Edwards MH, Dennison EM, Cooper C. Epidemiology and burden of osteoarthritis. Br Med Bull. 2013;105:185-99. doi: 10.1093/bmb/lds038. Epub 2013 Jan 20. PMID 23337796
- [Result] Michael JW, Schluter-Brust KU, Eysel P. The epidemiology, etiology, diagnosis, and treatment of osteoarthritis of the knee. Dtsch Arztebl Int. 2010 Mar;107(9):152-62. doi: 10.3238/arztebl.2010.0152. Epub 2010 Mar 5. PMID 20305774